CLINICAL TRIAL: NCT07204873
Title: Evaluation of the LUSHA Digital Application for Children With ADHD (Attention Deficit Hyperactivity Disorder) Feasibility Study
Brief Title: Evaluation of the LUSHA Digital Application for Children With ADHD - Feasibility Study
Acronym: LUSHA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: DYGIE (France) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC24.0245
Record Dates: First submitted 2025-08-19; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Attention Deficit Disorder With or Without Hyperactivity (ADHD); Children
Keywords: Attention Deficit Disorder with or without Hyperactivity (ADHD); Digital application; Psychoeducation; Cognitive behavioral therapy (CBT); Familiy quality of life; Parenting skills training (Barkley program)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of LUSHA digital app (Experimental)
  Interventions: Other: LUSHA digital app

INTERVENTIONS:
Other: LUSHA digital app — Children with Attention Deficit Disorder with or without Hyperactivity (ADHD) and their parents will be asked to use LUSHA app during 3 months.

SUMMARY:
Attention Deficit Disorder with or without Hyperactivity (ADHD) is a neurodevelopmental disorder characterized by a triad of symptoms combining inattention, hyperactivity, and/or impulsivity. It causes developmental and functional disturbances (cognitive, behavioral, and emotional) that have a detrimental impact on the child's family, school, and/or social life. Treatment requires psychoeducation for the child and their parents, individual treatment for the child, and finally family treatment, particularly through specific parenting skills training programs (such as the Barkley program, 1997). It is sometimes necessary to combine this with medication (psychostimulants).

This care pathway can be complex to implement in practice, due to lack of regional actors (CMPPs, medical-psychological-educational centers) and a decrease in the number of child psychiatrists in hospital services.

Recently, digital applications enabling the digitization of the psychotherapeutic approach have been developed to complement and reinforce the care provided to these children, offering an immediately available non-pharmacological alternative.

LUSHA is a digital application (digital game) developed in collaboration with healthcare professionals. It aims to motivate the children to change their behavior and help parents to interact with them.

The goal of this observational study is to evaluate the adoption of LUSHA app by children with Attention deficit disorder with or without Hyperactivity (ADHD) and their parents :

* The primary objective of this study is to assess adherence/use of a digital application among children with ADHD and their parents over a period of 90 days
* The secondary objectives are to assess the clinical impact of the LUSHA digital application using validated questionnaires (i.e quality of life, behavioural, family functioning).

Participating children and their parents will be asked to use the LUSHA digital application during 3 months and to answer online surveys.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-12 years
* Already diagnosed with ADHD
* Consulting in a participating center
* No indication of treatment changes (no treatment or medication stabilized for 2 months)
* Family with a smartphone compatible with downloading the app
* Non-opposition of both parents and the child (if possible)

Exclusion Criteria:

* Parent under guardianship or deprived of liberty

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the use of the LUSHA app among children and their parents at 3 months. | 90 days
  Use is defined as a cumulative usage of more than 30 minutes per week on average within 3 months (90 days) of app installation.

SECONDARY OUTCOMES:
To evaluate the use of the LUSHA app by children and their parents at 1 and 2 months. | 30, 60 days
  Use is defined as a cumulative usage of more than 30 minutes per week on average within 30 and 60 days of app installation.
To evaluate the quality of life (familial impact) before/after using the app | Inclusion, 30, 60, 90 days
  Number and proportion of children with functional impairment identified by the WFIRS-P parent questionnaire (Weiss Functional Impairment Rating Scale - Parent report; CADDRA, 2011)
To evaluate the evolution of the 5 questions of the app | 7, 30, 60, 90 days
  Average rating of responses to each of the 5 questions in the app (questions are asked directly in the application). Each question is rated from 1 to 10.
To evaluate behavioral impact before/after using LUSHA app | Inclusion, 30, 60, 90 days
  Number and proportion of children with behavioral abnormalities identified by the SNAP IV questionnaire (average sub-scores and overall scores) completed by parents (Swanson, Nolan, and Pelham Questionnaire - Swanson et al., 1999)
To evaluate the quality of life as assessed by the child before/after using the app | Inclusion, 30, 60, 90 days
  Overall, physical health, and psychosocial health (emotional + social + academic) mean scores on the questionnaire (PedsQL™ 4.0) Pediatric Quality of Life Inventory Version 4.0 Parent and child version (Varni et al, 2003), pediatric quality of life inventory (Appendix 3)
Appropriation of the functionnalities of the app by children and parents | 30, 60, and 90 days
  Description of the number of validated routines, modules on emotion management, modules on the Barkley program
Association between the clinical presentation of children with ADHD and comorbidities and use of the LUSHA app | 90 days
  Measurement of associations between average weekly usage, number of validated routines, modules completed on emotion management, modules completed on the Barkley program, and scores obtained on various questionnaires (WFIRS, SNAP, PedsQL)
Association between appropriation of the various functionalities of the app by children and parents and the familial impact, behavioral impact, and quality of life as assessed by the child. | 90 days
  Measurement of associations between average weekly usage time, number of validated routines, modules completed on emotion management, modules completed on the Barkley program, and scores obtained on various questionnaires (WFIRS, SNAP, PedsQL)

CONTACTS AND LOCATIONS:
Overall Officials: BIOULAC Stéphanie, Pr, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - University Hospital, Grenoble, Grenoble
  - University Hospital, Montpellier, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided